CLINICAL TRIAL: NCT06228794
Title: The Prognostic Value of Circulating Plasma Cells Quantified by Multiparameter Flow Cytometry in Patients With Multiple Myeloma: a Prospective, Multicenter Clinical Trial
Brief Title: The Prognostic Value of CPCs Quantified by Flow Cytometry in Patients With Multiple Myeloma: a Prospective, Multicenter Clinical Trial
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chunyan Sun, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: UHCT230750
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Circulating plasma cells; Multiparameter flow cytometry; Prognosis; Disease monitoring
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Newly diagnosed multiple myeloma cohort: Participants who meet the multiple myeloma diagnostic criteria of IMWG are eligible.
  Interventions: Other: Peripheral blood test

INTERVENTIONS:
Other: Peripheral blood test — We will draw 2-5 mL of peripheral blood and utilize multiparameter flow cytometry to measure the level of circulating plasma cells.

SUMMARY:
This study aims to investigate the prognostic value of circulating plasma cells (CPCs) in patients with multiple myeloma and explore whether CPCs detection might be used in place of bone marrow aspiration for disease monitoring.

DETAILED DESCRIPTION:
Circulating plasma cells (CPCs) represents a phenotypic subset of bone marrow multiple myeloma (MM) cells, which would contribute to the progression and dissemination of the tumor. High-sensitivity techniques such as multiparameter flow cytometry provide a tool for better detection of CPCs; however, a clear threshold has not been identified. The primary objective of the current study is to identify an optimal threshold for CPCs quantified by 8-color flow cytometry (with antibodies to CD38, CD138, CD45, CD56, CD19, CD27 and cytoplasmic kappa and lambda immunoglobulin light chains) and determine the specific relationship between CPCs level and the prognosis of MM. In addition, the evaluation of CPCs at multiple time points will be performed to explore whether CPCs detection might be used in place of bone marrow aspiration for disease monitoring.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria.

* Newly diagnosed multiple myeloma patients.
* Patients without any previous anti-myeloma treatment.
* Age: 18-80years old (adult).
* No history of cancer.
* Informed consent.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria will not be included in the study.

* Received therapy for multiple myeloma.
* Patients diagnosed with monoclonal gammopathy of undetermined significance, smoldering myeloma, nonsecretory myeloma, plasma cell leukemia, amyloidosis, waldenstrom macroglobulinemia or POEMS.
* Imminent or emerging infection.
* Known to be seropositive for a history of HIV.
* A participant is a woman who is pregnant, breastfeeding, or planning to become pregnant while enrolled in this trial.
* Known or suspected of not being able to comply with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed multiple myeloma patients
Sampling Method: Non-Probability Sample
Enrollment: 458 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (PFS) | 2 years
  To evaluate if there is a correlation between high CPCs level and poor PFS.

SECONDARY OUTCOMES:
Rates and depth of response | 2 years
  To evaluate if there is a correlation between CPCs level and rates and depth of response (IMWG response criteria).
Overall survival (OS) | 2 years
  To evaluate if there is a correlation between high CPCs level and poor OS.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided